CLINICAL TRIAL: NCT05557149
Title: Development and Evaluation of a Virtual Reality Application for Eliciting Craving and Its Physiological Arousal in Cocaine Users
Brief Title: Virtual Reality Exposure and Respiratory Relaxation-Based Coping With Cocaine Craving in Cocaine Users
Acronym: RVCOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire de Psychologie des Cognitions (Other)
Collaborators: ICube Laboratory - Team IGG (Unknown); Ithaque Association (Unknown); University Hospitals of Strasbourg (Unknown); University Hospital, Strasbourg, France (Other); The French National Cancer Institute (Unknown); The French Institute for Public Health Research (Unknown)
Responsible Party: Principal Investigator, Thomas Lehoux, Ph.D. Candidate, Laboratoire de Psychologie des Cognitions
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RVCOC2021; AAC21-SPA-04 (Other Grant/Funding Number: The French Institute for Public Health Research & The French National Cancer Institute); 2021-A00242-39 (Other: French Agency for the Safety of Health Products (ANSM)); 21.02.14.82513 (Other: Research Ethic Committee (CPP) - Sud Méditerranée V)
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Virtual Reality Exposure Therapy; Cocaine Use Disorder
Keywords: Virtual Reality; Cocaine Craving; Cue Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutral VR (Sham Comparator): Ten minutes virtual reality exposure to neutral stimuli (e.g. neutral picture frames)
  Interventions: Device: Virtual Reality Exposure to Neutral Cues
- Cocaine VR (Experimental): Ten minutes virtual reality exposure to cocaine use-related stimuli (i.e. peers using cocaine, cocaine paraphernalia, cocaine use preparing, cocaine use, etc.)
  Interventions: Device: Virtual Reality Exposure to Cocaine-Related Cues
- Relaxation (Other): Ten minutes respiratory relaxation (eyes closed and sitted on a chair)
  Interventions: Behavioral: Respiratory Relaxation

INTERVENTIONS:
Device: Virtual Reality Exposure to Neutral Cues — Virtual reality exposure to neutral stimuli (360 degrees visual and audio immersion with Oculus Quest 2 virtual reality headset). Participants stay sitted on chair and can tilt, rotate and move forward and backward upper body members. No interaction with the investigator during the virtual reality immersion.
  Arms: Neutral VR
Behavioral: Respiratory Relaxation — Respiratory relaxation practise. No interaction with the investigator during the relaxation practise.
  Arms: Relaxation
Device: Virtual Reality Exposure to Cocaine-Related Cues — Virtual reality exposure to cocaine-related stimuli (360 degrees visual and audio immersion with Oculus Quest 2 virtual reality headset). Participants stay sitted on chair and can tilt, rotate and move forward and backward upper body members. No interaction with the investigator during the virtual reality immersion.
  Arms: Cocaine VR

SUMMARY:
Our study main objective is to test whether virtual reality exposure could elicit cocaine craving and its physiological arousal in cocaine users. Investigators aim to compare self-reported cocaine craving, self-efficacy to cope with craving and emotional states levels in 11 voluntary and adults cocaine users in 3 consecutive 10-mins conditions: Neutral VR (virtual reality exposure to neutral stimuli), Cocaine VR (virtual reality exposure to cocaine use-related stimuli) and Relaxation (respiratory relaxation).

ELIGIBILITY:
Inclusion Criteria:

- Cocaine use within the past 28 days

Exclusion Criteria:

* Actual manic or hypomanic episode (MINI, Lecrubier and al., 1998)
* Actual psychotic episode (MINI, Lecrubier and al., 1998)
* Actual high suicidal risk (MINI, Lecrubier and al., 1998)
* Being involved in incarceration procedure
* Medical risk for safety while physiological arousal (e.g. cardiac disease)
* Disability for performing virtual reality task (e.g. blindness or deafness)
* Significant motion sickness symptoms (SSQ pre-post total score ≥ 15, Bimberg et al., 2020)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Cocaine Craving Intensity | Immediatly after Neutral VR, Cocaine VR and Relaxation (10 mins between each measure)
  Change in self-reported cocaine craving intensity between 3 consecutive interventions: Neutral VR, Cocaine VR and Relaxation (CCQ-Brief total score, french version; Karila and al., 2011). CCQ-Brief total score varies from 10 to 70 (higher score suggesting higher craving intensity).

SECONDARY OUTCOMES:
Self-Efficacy to Cope with Cocaine Craving without Using | Immediatly after Neutral VR, Cocaine VR and Relaxation (10 mins between each measure)
  Change in self-reported efficacy level to cope with cocaine craving without using between 3 consecutive interventions: Neutral VR, Cocaine VR and Relaxation (DTCQ-8 total score, original version translated in french; Sklar and Turner, 1999). DTCQ-8 total score varies from 0 to 800 (higher score suggesting higher self-efficacy to cope with cocaine craving without using).
Negative Emotional States | Immediatly after Neutral VR, Cocaine VR and Relaxation (10 mins between each measure)
  Change in negative emotional states level between 3 consecutive interventions: Neutral VR, Cocaine VR and Relaxation (BMIS negative emotional states total score, adapted version translated in french Mayer et al., 1988). BMIS negative emotional states total score varies from 0 to 21 (higher score suggesting higher negative emotional states).
Positive Emotional States | Immediatly after Neutral VR, Cocaine VR and Relaxation (10 mins between each measure)
  Change in positive emotinal states level between 3 consecutive interventions: Neutral VR, Cocaine VR and Relaxation (BMIS positive emotional states total score, adapted version translated in french Mayer et al., 1988). BMIS positive emotional states total score varies from 0 to 9 (higher score suggesting higher positive emotional states).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lehoux, Ph.D. Candidate, Principal Investigator — Laboratoire de Psychologie des Cognitions (Strasbourg University)
Locations (1):
- Laboratoire de Psychologie des Cognitions (Strasbourg University), Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: No